CLINICAL TRIAL: NCT02667431
Title: Cancer of the Uterus and Treatment of Stress Urinary Incontinence
Acronym: CUTI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: University of Alabama at Birmingham (Other); Hartford Hospital (Other)
Responsible Party: Principal Investigator, Katina Robison, MD, Women and Infants Hospital of Rhode Island
Other Study IDs: 823303-1
Record Dates: First submitted 2015-12-02; First posted 2016-01-29 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Endometrial Cancer; Stress Urinary Incontinence
Keywords: SUI
MeSH Terms: conditions — Endometrial Neoplasms; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Concurrent treatment of endometrial cancer and SUI may improve QOL, emotional and physical health and decrease costs for both patients and the health care system. At the time of endometrial cancer diagnosis, not only are women evaluated by a gynecologist and/or a gynecologic oncologist, but the majority will undergo surgery within weeks of their diagnosis. Thus, urinary incontinence could easily be identified, a referral made, and concurrent surgery performed. This would spare the patient two surgeries, decrease the emotional distress associated with SUI symptoms, decrease the costs associated with SUI for the patient and possibly improve overall quality of life. The proposed study will compare the quality of life and clinical outcomes among women with endometrial cancer and SUI that have concurrent surgery to women that do not have concurrent surgery. The findings of our proposed research will provide valuable information necessary for woman and clinicians to make decisions regarding the treatment of SUI, including evidence regarding the risks and benefits of performing concurrent endometrial cancer and SUI surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women will be eligible if they have:

  1. clinical stage 1 or 2 (disease confined to the uterus) endometrial carcinoma or complex atypical hyperplasia
  2. answer yes to one screening question: "Do you ever leak urine when you cough, sneeze, jump or laugh?" We will include women with complex atypical hyperplasia (CAH) because 40% of these women will have an endometrial cancer identified at the time of surgery and the risk factors are the same for CAH as they are for clinical stage 1 and 2 endometrial cancers

Exclusion Criteria:

* Women will be excluded if they have

  1. clinical stage 3 and 4 endometrial cancer
  2. prior pelvic radiation therapy
  3. vesicovaginal fistula
  4. urethrovaginal fistula.
* We are excluding women with vesicovaginal fistula or urethrovaginal fistula due to the risk of infection when placing a midurethral sling.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed complex atypical hyperplasia or clinical stage 1 or 2 endometrial cancer based on physical exam and/or imaging will be approached.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Pre-op to 12 month post-op
  The purpose of this study is to compare quality of life among women with endometrial cancer and SUI who undergo SUI and endometrial cancer surgery simultaneously to women that do not.
Sexual Function will be measured using the female sexual function index (FSFI) | Pre-op to 12 month post-op
  Compare the sexual function of women with endometrial cancer and SUI who have concurrent surgery to women who have cancer surgery only. Sexual function will be measured using the female sexual function index (FSFI). It is a 19-item instrument assessing 6 domains of sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain.
Clinical Outcomes- Time to Surgery | Enrollment to Day of Surgery
  Compare the clinical outcomes of women with endometrial cancer and SUI who have concurrent surgery to women who have cancer surgery only, by measuring time to surgery (ie: number of days) using hospital records. The estimated time to surgery will be assessed up to 12 weeks, measuring from initial date of enrollment to date of documented surgery date.
Clinical Outcomes- Surgical Outcomes | Pre-op to 12 month post-op
  Compare the clinical outcomes of women with endometrial cancer and SUI who have concurrent surgery to women who have cancer surgery only by examining surgical outcomes such as intra op injuries or complications using hospital records.
Clinical Outcomes- Post-Operative Complications | Pre-op to 12 month post-op
  Compare the clinical outcomes of women with endometrial cancer and SUI who have concurrent surgery to women who have cancer surgery only by examining Post-Operative complications. We will document any treatment-related adverse events as assessed by CTCAE v4.0. We will use hospital records.

SECONDARY OUTCOMES:
Sling Complications | Pre-op to 12 month post-op
  Compare the rate of midurethral sling complications among women who received radiation after sling placement to women who did not receive radiation using hospital records.
Post- Operative Pain | Day 1 in hospital after surgery
  We will also measure post-operative pain, using the modified Brief Pain Inventory (BPI) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robison K, Wohlrab K, Howe CJ, Richter HE, Sung V, Bevis KS, Luis C, McCourt C, Lowder J, Occhino J, Glaser G, Lokich E, Dunivan G, Brown A, Tunitsky-Bitton E, Wethington S, Chen CCG, Rahn D, Carlson M, Cram R, Raker C, Clark MA. Endometrial Cancer Surgery With or Without Concomitant Stress Urinary Incontinence Surgery. Obstet Gynecol. 2023 Apr 1;141(4):642-652. doi: 10.1097/AOG.0000000000005059. Epub 2023 Mar 9. PMID 36897162